CLINICAL TRIAL: NCT03979781
Title: Personalized Antiplatelet Secondary Stroke PRevenTion (PASSPoRT). A Randomized, Phase II, Open Label, Trial in High Risk Transient Ischemic Attack (TIA) and Ischemic Stroke Survivors Age 18 Years and Older
Brief Title: Personalized Antiplatelet Secondary Stroke PRevenTion
Acronym: PASSPoRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1158092
Record Dates: First submitted 2019-03-18; First posted 2019-06-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Ischemic Stroke; TIA
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Intervention group
  Interventions: Drug: tailored antiplatelet selection
- Control Group (Active Comparator): Standard of Care group
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: tailored antiplatelet selection — antiplatelet selection guided by platelet function phenotype and/or key pharmacogene genotypes
  Arms: Treatment Group
Drug: standard of care — antiplatelet selection using standard of care
  Arms: Control Group

SUMMARY:
This is a descriptive study designed to evaluate the safety and feasibility of a precision medicine approach to antiplatelet selection for secondary stroke prevention.

DETAILED DESCRIPTION:
Subjects meeting inclusion/exclusion criteria will be randomly assigned to: (1) the treatment group where antiplatelet medications will be selected using platelet function phenotype and/or key pharmacogene genotypes (2) the control group where participants will receive standard care for antiplatelet therapy (without knowledge of phenotype or genotype).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Meet criteria for a mild or moderate ischemic stroke or high-risk TIA
* Ability to randomize within 30 hours of stroke symptom onset/last seen normal time

Exclusion Criteria:

* Evidence of new or prior non-traumatic intracerebral hemorrhage, subarachnoid hemorrhage, or subdural hemorrhage on initial head CT
* Evidence of a central nervous system tumor, abscess, intracranial aneurysm or vascular/structural malformation, or any neuro-inflammatory, neuro-infectious, or neurodegenerative disorder on neuroimaging or exam that could confound a participant's functional outcome
* Isolated or pure sensory symptoms (e.g., numbness), visual changes, or "dizziness"/vertigo without evidence of acute ischemic stroke on baseline head CT or MRI.
* Qualifying ischemic event is believed to be iatrogenic or procedure related
* Required to take a specific antiplatelet medication for an indication other than ischemic stroke during the study period that would prevent the investigator from following the study algorithm
* Etiology of qualifying ischemic event is known to be cardioembolic
* High likelihood that anticoagulation will be needed during the study period.
* High likelihood that carotid endarterectomy or carotid stenting will occur during the period of the study.
* Pre-stroke modified Rankin scale (mRS) score ≥ 3
* Evidence of frailty
* Contraindication to aspirin, clopidogrel, Aggrenox®, or ticagrelor
* Known allergy or hypersensitivity that would prevent the investigator from following the study algorithm
* Any history of moderate to severe drug-induced adverse events
* Renal insufficiency or history of kidney transplant
* Hepatic impairment, international normalized ratio (INR) > 1.5, physical manifestations of liver disease, or history of liver transplant
* Class II, III, or IV New York Heart Association (NYHA) functional heart failure
* Any history of bradycardia without pacemaker placement
* Active obstructive lung disease
* Any active hematologic disorder
* Active bleeding diathesis
* Any systemic hemorrhage or GI bleed in the 3 months prior to the qualifying stroke
* Active peptic ulcer disease
* Women who self-report that they are pregnant or breastfeeding
* Active alcohol or substance abuse or dependence
* Inability or failure to provide informed consent.
* Inability of the patient to adhere to study procedures and/or follow-up, in the opinion of the investigative team
* Inability to swallow oral medications
* Not willing or able to discontinue prohibited concomitant medications
* Ongoing participation in another non-observational clinical study
* Life expectancy < 1 year, in the opinion of the investigative team

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment and Platelet Reactivity | 90 days
  ability to recruit participants and achieve platelet reactivity target using platelet function assays
Safety - Bleeding Complications | 90 days
  bleeding questionnaire
Safety - Bleeding Complications | 1 year
  bleeding questionnaire

SECONDARY OUTCOMES:
Patient-centered Outcomes - Satisfaction | 90 days
  consumer assessment of healthcare providers and systems
Patient-centered Outcomes - Satisfaction | 1 year
  consumer assessment of healthcare providers and systems

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Albright, PhD, DO, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No